CLINICAL TRIAL: NCT01814735
Title: Substituting Brown Rice For White Rice: Effect On Diabetes Risk Factors In India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Madras Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Frank B. Hu, Professor of Nutrition and Epidemiology, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: R03TW008726-01 (NIH)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brown rice (Experimental): Brown Rice
  Interventions: Other: Brown rice; Other: White rice
- White rice (Active Comparator): White rice
  Interventions: Other: Brown rice; Other: White rice

INTERVENTIONS:
Other: Brown rice
Other: White rice

SUMMARY:
Currently, India has the largest absolute number of people with diabetes in the world, and evidence indicates that consumption of whole-grains can decrease diabetes by improving glycemic control. Our study will evaluate the efficacy of substituting brown rice, a whole-grain, for white rice in Chennai, India, on biomarkers of diabetes risk. The ultimate goal of this research is to provide data for use in designing a global dietary intervention study aimed at reducing diabetes risk through simple, culturally appropriate, feasible and sustainable dietary changes.

DETAILED DESCRIPTION:
Currently, India has the largest absolute number of people with diabetes in the world and the escalation in diabetes incidence is occurring as global free trade continues to fuel rapid economic and nutrition transitions, especially in urban settings. These transitions are accompanied by a shift in dietary consumption towards more highly refined carbohydrates, fats, and animal products. Evidence indicates that consumption of whole-grains can decrease diabetes by improving glycemic control. The proposed proof-of-concept trial herein will evaluate the efficacy of substituting brown rice, a whole-grain, for white rice in Chennai, India, on biomarkers of diabetes risk and also will obtain glycemic index values of local rice and other staples. The long-term goal is to develop a multi-center nutritional-intervention in India, China, Africa and Latin America to create sustainable diabetes prevention strategies through improving carbohydrate quality. The investigators propose to conduct a 4-month randomized parallel-group intervention trial to evaluate the effects of substitution of brown rice for white rice in two meals per day six days per week on biomarkers for diabetes risk among adults in Chennai, India who are at high risk for the development of diabetes. The first aim of this research is to determine the glycemic index of different local rice varieties (brown, red, and fully polished white) and preparations (regular or parboiled). The second aim is to determine the effects of brown rice substitution on fasting biomarker measurements of glucose metabolism (i.e., glucose, insulin, hemoglobin A1c, homeostasis model assessment for insulin resistance), dyslipidemia (i.e., triglycerides, total cholesterol, LDL- cholesterol, and HDL-cholesterol), and inflammation (i.e., C-reactive protein). This trial will also demonstrate the feasibility and cultural appropriateness of this type of intervention in the local environment to which results may be translated in the future. This study will have important implications for policy and help local governments develop national nutrition strategies for diabetes prevention such as wide- spread education campaigns about the health benefits of whole-grains, and school lunch programs which serve whole-grains. Such policies could also encourage ministries of agriculture to support production of whole grains, thereby improving accessibility and regulate costs. This work is intended to be part of a larger global initiative to identify local, feasible and sustainable dietary interventions to reduce diabetes risk in countries experiencing epidemiologic transition by improving the carbohydrate quality of staple foods. Initiatives have already been launched by our group in China, and are planned for Tanzania, Nigeria, Puerto Rico and Mexico. PUBLIC HEALTH RELEVANCE: Currently, India has the largest absolute number of people with diabetes in the world, and evidence indicates that consumption of whole-grains can decrease diabetes by improving glycemic control. Our study will evaluate the efficacy of substituting brown rice, a whole-grain, for white rice in Chennai, India, on biomarkers of diabetes risk. The ultimate goal of this research is to provide data for use in designing a global dietary intervention study aimed at reducing diabetes risk through simple, culturally appropriate, feasible and sustainable dietary changes.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index > 23kg/m2 (India-specific BMI cutpoint for overweight)
2. Waist circumference ≥ 90cm if male and ≥ 80cm if female (India-specific cutpoints for abdominal adiposity)
3. Daily rice consumption (≥200grams/day, > ~2cups/day) as determined by responses to the screening questionnaire

Exclusion Criteria:

1. Self-report of any condition/illness that may affect the study outcomes or would make participation potentially harmful, including diabetes, severe kidney disease, cardiovascular disease (coronary artery disease, peripheral vascular disease), history of stroke, cancer, severe psychological disorders (schizophrenia, dementia), or hypothyroidism, as ascertained by a detailed medical history.
2. No plans to relocate in the next year.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in fasting blood glucose, lipids, and blood pressure | 4 months

SECONDARY OUTCOMES:
Feasibility and cultural appropriateness | 1 year
  This trial will also demonstrate the feasibility and cultural appropriateness of this type of intervention in the local environment to which results may be translated in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Madras Diabetes Research Foundation, Chennai, India